CLINICAL TRIAL: NCT00901758
Title: Intravenous (IV) Nitroglycerin for Versions in Multiparous Women
Acronym: INVERT (02)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Dr B Allan, Department of Obstetrics and Gynecology, Rockyview General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INVERT-02; CHREB #16682
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Breech Presentation; Pregnancy Complication
MeSH Terms: conditions — Breech Presentation; Pregnancy Complications | interventions — Nitroglycerin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Placebo solution was normal saline. After an initial 1mL dose, further doses could be given in 1-3mL increments until uterine relaxation was achieved, or up to a recommended maximum of 10mL.
  Interventions: Drug: Normal saline
- 1 (Active Comparator): Treatment solution consisted of 100micrograms/mL of nitroglycerin. After an initial 1mL dose, further doses could be given in 1-3mL increments until uterine relaxation was achieved, or up to a recommended maximum of 10mL.
  Interventions: Drug: IV Nitroglycerin

INTERVENTIONS:
Drug: IV Nitroglycerin — IV injection, initial does of 1mL, with further doses of 1-3mL, up to a recommended maximum of 10mL.
  Arms: 1
Drug: Normal saline — IV injection, initial does of 1mL, with further doses of 1-3mL, up to a recommended maximum of 10mL
  Arms: 2

SUMMARY:
Breech presentations (where a baby presents with feet or bottom down) have an increased risk of perinatal and neonatal complications, and are usually delivered by cesarean section. As an alternative, so that the baby can be delivered vaginally, an attempt can be made to turn the baby so that it is head down: this manoeuvre is called an external cephalic version (ECV).

Drugs that relax the uterus (tocolytic agents) are sometimes used to help improve ECV success rates. Nitroglycerin is a tocolytic agent, but intravenous nitroglycerin has not been tested as an agent to help ECV. There is some suggestion that nitroglycerin may be more helpful in women who have not previously been pregnant (nulliparous women) than in women who have been pregnant more than once (multiparous women), and so we have planned two trials.

This study is designed to answer the following questions for multiparous women:

Will administration of IV nitroglycerin for uterine relaxation improve ECV success rates? Will an increase in ECV success result in a decreased cesarean section rate?

ELIGIBILITY:
Inclusion Criteria:

* any non-cephalic presentation
* singleton pregnancy
* >/= 37 weeks gestational age
* normal amniotic fluid volume
* reassuring fetal heart rate

Exclusion Criteria:

* labor
* ruptured membranes
* history of third trimester bleeding
* any pre-existing uterine scar
* pregnancy induced hypertension and gestational diabetes
* oligohydramnios and polyhydramnios
* intrauterine growth restriction or macrosomia
* hypotension or any serious medical illness
* inability to comprehend consent form

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-03; Primary Completion 2006-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Success of ECV (if fetus turned from Breech to cephalic) at end of ECV procedure | Recorded at the end of ECV attempt

SECONDARY OUTCOMES:
Success of ECV (ie fetus in cephalic presentation) recorded at time of delivery | Recorded at time of birth
Mode of delivery | Recorded at time of birth
Maternal side effects and adverse events | Recorded until date of birth (up to 3 weeks' duration).

CONTACTS AND LOCATIONS:
Overall Officials: Bruce B Allan, MD PhD, Principal Investigator — Calgary Health Region
Locations (3):
- Canada (3):
  - Foothills Medical Centre, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - Rockyview Hospital, Calgary, Alberta

REFERENCES:
- [Result] Hilton J, Allan B, Swaby C, Wah R, Jarrell J, Wood S, Ross S, Tran Q. Intravenous nitroglycerin for external cephalic version: a randomized controlled trial. Obstet Gynecol. 2009 Sep;114(3):560-567. doi: 10.1097/AOG.0b013e3181b05a19. PMID 19701035